CLINICAL TRIAL: NCT04947124
Title: Masked, Randomized, Single-site, Crossover Study to Determine the Safety and Tolerability of 2 Concentrations of QLS-101 Dosed for 14 Days in Adult Subjects With Sturge-Weber Syndrome (SWS)-Related Glaucoma Due to Elevated Episcleral Venous Pressure (EVP)
Brief Title: A Study to Determine the Safety and Tolerability of 2 Concentrations of QLS-101
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Qlaris Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: QC-203
Record Dates: First submitted 2021-06-08; First posted 2021-07-01 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Sturge-Weber Syndrome (SWS); Glaucoma; Glaucoma Congenital; Ocular Hypertension
Keywords: Sturge-Weber Syndrome; Glaucoma; Elevated Intraocular pressure (IOP)
MeSH Terms: conditions — Sturge-Weber Syndrome; Glaucoma; Hydrophthalmos; Ocular Hypertension

STUDY DESIGN:
Intervention Model Description: Patients take 2 different doses of investigational product at distinct treatment periods. Dose is masked.
Who Masked: Participant, Investigator
Masking Description: Masked investigational product labeling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1% QLS-101 (Experimental): dosed once a day for 14 days as either first or second dosing period per randomization
  Interventions: Drug: QLS-101ophthalmic solution 1%
- 2% QLS-101 (Experimental): dosed once a day for 14 as either first or second dosing period per randomization
  Interventions: Drug: QLS-101ophthalmic solution 2%

INTERVENTIONS:
Drug: QLS-101ophthalmic solution 1% — QLS-101ophthalmic solution 1.0%
  Other Names: QLS-101
  Arms: 1% QLS-101
Drug: QLS-101ophthalmic solution 2% — QLS-101ophthalmic solution 2.0%
  Other Names: QLS-101
  Arms: 2% QLS-101

SUMMARY:
Safety and tolerability study of 2 concentrations of QLS-101 for adult subjects with Sturge Weber Syndrome (SWS)-related glaucoma due to elevated episcleral venous pressure (EVP).

DETAILED DESCRIPTION:
Masked, randomized, single site, crossover study to compare 2 concentrations of QLS-101. Subjects will be randomized to one of 2 concentrations of QLS-101 for the first 14 days of daily dosing, and after a 14-day washout period they will be crossed over to the other concentration for another 14 days of daily dosing. Dose assignment is masked to patient and investigator.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with SWS.
* Elevated intraocular pressure (IOP)
* Willing to continue current dosing regimen of IOP-lowering medications
* Willing to refrain from contact lens use in the study eye.

Exclusion Criteria:

* IOP with variability of > 4 mm Hg
* Expected to undergo IOP-lowering surgery
* Incisional or laser surgery of any type
* Ocular infection, inflammation, clinically significant blepharitis or conjunctivitis
* A history of herpes simplex keratitis in either eye.
* History of or active clinically significant ocular disease
* Use of topical ocular corticosteroids in the 6 weeks prior to Visit 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Ocular adverse events (AEs) | 56 days, including a 14-day washout
  Standard safety endpoint, ocular AEs, (including elevated IOP)
Visual acuity | 56 days, including a 14-day washout
  Standard safety endpoint, best corrected visual acuity, Snellen score, change from baseline
Enhance depth imaging optical coherence tomography (EDI-OCT) | 56 days, including a 14-day washout
  Standard safety endpoint, EDI-OCT, corneal thickness
Slit lamp exam | 56 days, including a 14-day washout
  Standard safety endpoint, slit lamp exam, abnormalities, changes from baseline
Dilated fundus exam | 56 days, including a 14-day washout
  Fundus exam, abnormalities, changes from baseline

SECONDARY OUTCOMES:
Ocular hypotensive efficacy | 14 days after each dosing timepoint is completed
  Mean change in IOP from baseline following 14 days dosing

CONTACTS AND LOCATIONS:
Overall Officials: B. Wirostko, M.D., Study Director — Qlaris Bio, Inc.
Locations (1):
- Duke Eye Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Qlaris Bio website, pipeline page — https://qlaris.bio